CLINICAL TRIAL: NCT00210769
Title: Open-label Extension of A Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel-Group, Dose-Response Study to Evaluate the Efficacy and Safety of 2 Fixed Dosages of Extended Release OROS� Paliperidone (6 and 12 mg/Day) and Olanzapine (10 mg/Day), in Patients With Schizophrenia
Brief Title: A Study of the Long-term Safety and Tolerability and the Long-term Effectiveness of Extended-release Oral Paliperidone in Patients Diagnosed With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004426
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; extended release; oral administration; antipsychotic agents; dementia praecox; mental disorders; paliperidone; PANSS
MeSH Terms: conditions — Schizophrenia; Mental Disorders

INTERVENTIONS:
Drug: paliperidone ER Oros

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability and the maintenance of effectiveness of a slow, extended-release oral formulation of paliperidone administered once daily to patients diagnosed with schizophrenia.

DETAILED DESCRIPTION:
The controlled rate of drug delivery provided by the extended-release oral formulation of paliperidone may provide improved effectiveness and a reduced risk of certain adverse effects in patients with schizophrenia, by avoiding peaks and troughs of drug levels in the blood. This could in turn provide an improved quality of life and overall functioning for patients.

This open-label study is an extension of a 6-week randomized, double-blind, parallel-group study in which the effectiveness and safety of 4 different oral treatments administered once daily are compared in patients with schizophrenia: paliperidone 6 or 12 milligrams (mg), olanzapine 10 mg (an approved treatment for schizophrenia), or placebo. Following the double-blind treatment phase, eligible patients may enter this 52-week open-label extension with slow, extended-release paliperidone (with no comparison treatments). In the open-label extension, all patients, regardless of their randomized treatment in the double-blind phase, will begin on extended-release paliperidone 9 mg once daily. Thereafter, patients will be maintained on a flexible dosage of extended-release paliperidone throughout the 52-week study. The dosage may be increased or decreased within this range in accordance with the clinical judgment of the investigator, based on observations of patient response and tolerability. Because flexible dosing more closely mimics clinical practice, this design may provide more clinically relevant findings in the open-label setting.The final visit in the double-blind phase may serve as the initial visit for the open-label extension. Study visits will occur at Day 4 and then weekly for the first 4 weeks (Weeks 1, 2, 3, and 4) and then every 4 weeks through Week 52 or until early termination. Evaluations of the safety and effectiveness of extended-release paliperidone treatment will be performed at scheduled times throughout the open-label extension. Flexible dosage (3, 6, 9, or 12 milligrams (mg)) extended-release paliperidone tablets administered orally once daily for 52 weeks, following a 6-week double-blind study in which patients receive fixed oral doses of 6 mg or 12 mg extended-release paliperidone or olanzapine 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* As for the double-blind study, a diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV)
* experiencing an acute episode of schizophrenia at time of screening for the double-blind study, with a total PANSS score of 70 to 120
* completed the double-blind study or discontinued after at least 21 days of double-blind treatment because of lack of efficacy
* for female patients of childbearing potential, agreement to continue to use an acceptable form of contraception throughout the open-label extension, with a negative urine pregnancy test at open-label baseline.

Exclusion Criteria:

* As for the double-blind study, a DSM-IV axis I diagnosis other than schizophrenia
* a DSM-IV diagnosis of substance dependence within 6 months prior to screening for the double-blind study
* considered by the investigator to be at significant risk for suicidal or violent behavior during the open-label study
* received an injection of a depot antipsychotic since entry into the double-blind study
* a woman who has become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2004-01; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Standard safety evaluations, and monitoring of extrapyramidal symptoms (tardive dyskinesia, akathisia) by the Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Rating Scale (BARS), and Simpson Angus Scale (SAS), throughout the long-term study.

SECONDARY OUTCOMES:
Assessment of long-term effectiveness by the Positive and Negative Syndrome Scale (PANSS), Clinical Global Impression Scale - Severity (CGI-S), Personal and Social Performance Scale (PSP), and Schizophrenia Quality of Life Scale, Revision 4 (SQLS-R4).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Kozma C, Dirani R, Canuso C, Mao L. Change in employment status over 52 weeks in patients with schizophrenia: an observational study. Curr Med Res Opin. 2011 Feb;27(2):327-33. doi: 10.1185/03007995.2010.541431. Epub 2010 Dec 15. PMID 21155708
- See also: A study of the long-term safety and tolerability and the long-term effectiveness of extended-release oral paliperidone in patients diagnosed with schizophrenia. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=595&filename=CR004426_CSR.pdf